CLINICAL TRIAL: NCT02035514
Title: Phase I-II Clinical Trial With Autologous Bone Marrow Derived Mesenchymal Stem Cells for the Therapy of Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Cristina Ramo, Phase I-II clinical trial with autologous bone marrow derived mesenchymal stem cells for the therapy of mutiple sclerosis., Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CELLTRiMS; 2010-024081-21 (EudraCT Number)
Record Dates: First submitted 2013-12-17; First posted 2014-01-14 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: multiple sclerosis; mesenchymal stem cells; autologous transplantation; MRI efficacy; clinical safety
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): A single infusion of up to 1 million cells per Kg of autologous MSC stem cells vs placebo. The treatment will be on day 0 and placebo on month 6.
  Interventions: Biological: Bone marrow autologous mesenchymal stem cells transplantation
- Arm 2 (Experimental): A single infusion of up to 1 million cells per Kg of autologous MSC stem cells vs placebo. The treatment will be on month 6 and placebo on day 0.
  Interventions: Biological: Bone marrow autologous mesenchymal stem cells transplantation

INTERVENTIONS:
Biological: Bone marrow autologous mesenchymal stem cells transplantation

SUMMARY:
Immunomodulatory therapies to treat the relapsing-remitting phase of multiple sclerosis (MS) are designed to ameliorate the inflammatory processes that mediate the damage to the central nervous system (CNS) and to delay progression of the disease. To date, there is no effective means to stop the progression of disease and induce remyelination. Adult stem cells therapy show great promise and is rapidly developing as alternative therapeutic strategy. We propose the use of bone marrow-derived autologous Mesenchymal (BM-MSC) Stem Cells transplantation to treat patients with relapsing-remitting MS (RRMS), despite immunomodulatory therapy. Taking advantage of the potential that MSC possess strong immunomodulatory properties thought to play a role in the maintenance of peripheral tolerance and in the control of autoimmunity and that may stimulate repair and regeneration of lesions, we plan a trial of a single injection of autologous BM-MSC into eight patients. First, we aim to assess the feasibility, safety and tolerability of autologous MSC therapy in RRMS. Second, we plan to evaluate the effects of BM-MSC transplantation on MS disease activity by clinical, neurophysiological, immunological and imaging assessments. Autologous MSC will be obtained from bone marrow aspirates, purified by culture and characterized by surface antigen expression. A single dose of autologous BM-MSC will be injected intravenously. Clinical, neurological and immunological assessments will be scheduled at baseline (before BM-MSC transplantation) at 1, 3, and 6 months after transplant. The imaging will be performed at 3 and 6 months after transplant. Proposed trial will enable us to ascertain whether autologous BM-MSC transplantation is a feasible and safe procedure, and whether BM-MSC can establish an environment of immune tolerance and through the local production of neurotrophic/growth factors, might induce neuroprotection and improvement in CNS function.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, demyelinating disease of the CNS. Onset typically occurs in early adulthood. Patients present with intermittent symptoms that are partially reversible; this form is termed relapsing-remitting (RRMS). Over time, most patients develop secondary-progressive MS (SPMS) which manifests as irreversible and gradual neurological impairments that often progress without acute relapses. Beta-interferons or glatiramer acetate represents the first line therapeutic option for RRMS. Clinical trials confirm that show partial efficacy, though they do not prevent the onset of secondary progression. SPMS, is the consequence of axonal loss and neurodegeneration and no current therapy has been effective. Stem cell therapy show great promise and is rapidly developing as alternative therapeutic strategy. Clinical indications for adult stem cells, which can be safely harvested and normally behave well without formation of tumours, are rapidly increasing. The majority of human stem cell trials have focused on clinical applications for haematopoietic stem cells (HSC), mesenchymal stem cells (MSC), or both, which can be easily obtained in clinically sufficient numbers from peripheral blood, bone marrow, adipose tissue, or umbilical cord blood and placenta. MSC can readily be isolated from a small sample of bone marrow and rapidly expanded so as to generate large numbers of cells for autologous therapies. When administered intravenously have an immune suppressive effect that can ameliorate animal autoimmune diseases. MSC transplantation significantly improves clinical outcome in experimental allergic encephalitis (EAE), the animal model of MS. When intravenously injected, MSC may migrate to inflammatory brain lesions and promote survival of brain-resident cells. Several disease models demonstrate axonal neuroprotection following MSC therapy, with some evidence that this is potentially mediated through the production of neurotrophic/growth factors, and/or immunomodulatory effects of MSC. For that reasons, MSC have become the focus of research as a potential cell therapy for inducing neuroprotection in human neurodegenerative diseases such as MS.

A growing body of literature confirms the therapeutic MSC biological properties, and provide a plausible mechanism of action to guide clinical trial design with a number of phase I/II trials in MS patients now underway. Experimental clinical trials in MS are being considered or have recently been initiated by several research groups, which are testing the therapeutic potential of different sources of MSC. Learning from previous clinical studies, and taking advantage of the potential that adult BM-MSC may stimulate repair and remyelination, to plan a clinical trial in patients with inflammatory MS seems reasonable. We propose a safety trial of a single intravenous injection of autologous bone marrow-derived MSC into 8 subjects with RRMS. The trial proposed here will enable us to ascertain whether autologous BM-MSC transplantation is a safe procedure, and whether BM-MSC therapy during the relapsing-remitting phase of MS can establish a immunomodulatory and regenerative microenvironment and reverse neurological disability in RRMS patients.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS (RRMS) patients
* Age 18-50 years
* Disease duration >= 2 and <= 10 years
* EDSS: 3.0 - 6.5
* 1) Patients who do not wish to be subjected to approved immunomodulatory treatments (interferon beta and acetato de glatiramer) 2) Patients who have tried and had to withdraw within a year due to adverse events 3) Patients who have not responded to them after at least 1 year of continuous treatment. Lack of response is considered one or more of the following

  * >= 1 moderate-severe relapses in past 12 months
  * >= 2 moderate-severe relapses in past 24 months
  * >= 1 Gadolinium enhancing lesions in a MRI performed in previous 12 months

Relapse:

* Mild: Increase of < 1 EDSS point
* Moderate: Increase of >= 1 EDSS point (if baseline EDSS 3.0-5.0) or 0.5 EDSS points (if baseline EDSS >= 5.5)
* Severe: Increase of >=3 EDSS point
* Social, mental and physical ability to communicate with physicians and to understand the requirements of the protocol
* Has given informed consent to participate in the study

Exclusion Criteria:

* RRMS not fulfilling inclusion criteria
* SPMS or PPMSTreatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
* Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
* Treatment with interferon-beta or glatiramer acetate within the 30 days prior to randomization
* Treatment with corticosteroids within the 30 days prior to randomization
* Relapse occurred during the 60 days prior to randomization
* History of cancer or clinical or laboratory results indicative of severe systemic diseases, including infection for HIV, Hepatitis B or C
* Pregnancy or risk of pregnancy/ lactation
* Current treatment with an investigational therapy
* Inability to give written informed consent in accordance with research ethics board guidelines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in safety | Baseline, month 12
  * Physical examination, vital signs (HR, RR, BP, axillary temp), analytical results (biochemistry, hematology,) electrocardiographic monitoring, pulse oximetry and adverse events.
  * Clinical worsening both new relapses or disability measured by Expanded Disability Status Scale (EDSS), until the end of the study.
Change from baseline in effectiveness by MRI | Baseline, month 6
  - Cumulative number of MRI Gd-enhancing lesions (3 and 6 months post-treatment).

SECONDARY OUTCOMES:
Feasibility | month 12
  - Availability of a viable product that allows the treatment, checking whether the procedures can be performed as indicated in protocol.
Change from baseline in effectiveness by MRI | baseline, month 3
  - Cumulative number of lesions visualized on T2 sequence (3 and 6 months post-treatment).
Change in clinical efficacy | baseline, month 1
  * EDSS score at months 1
  * Multiple Sclerosis Functional Composite (MSFC) scale at months 1
Change in Quality of life | Baseline, month 6 post-treatment
  - Multiple Sclerosis Quality of Life (MSQOL-54)
Immunology | baseline, month 6 post-treatment
  * Dosing of G, A and M immunoglobulins, and complement factors C3 and C4
  * Determination of lymphocyte subpopulations using cell surface staining and flow cytometry analysis. T lymphocyte subpopulations (CD4 and CD8), B lymphocytes, NK cells, dendritic and T regulatory cells will be analyzed
  * Quantification in serum by "Cytometricbeadarray" (CBA) and subsequent flow cytometry: IL-2, 4, 6, interferon (IFN) IFN-γ, interleukin (IL) IL-10, tumor necrosis factor (TNF) TNF-α or by ELISA: T-cell growth factor (TGF) TGF-β and IL-17.
Axonal effect | baseline, month 6
  - Optical coherence tomography (OCT)
Change from baseline in effectiveness by MRI | baseline, month 6
  - Cumulative number of lesions visualized on T2 sequence (3 and 6 months post-treatment).
Change in clinical efficacy | baseline, month 3
  * EDSS score at months 3
  * MSFC scale at months 3
Change in clinical efficacy | baseline, month 6 post-treatment
  * EDSS score at month 6 post-treatment
  * MSFC scale at month 6 post-treatment
  * Frequency of relapses 6 months post-treatment
  * Proportion of patients free of relapses 6 months post-treatment,
  * Number of relapses requiring corticosteroid treatment 6 months post-treatment
  * Time to first relapse from the baseline
Change in Quality of life | baseline, month 1
  - MSQOL-54
Change in Quality of life | baseline, month 3
  - MSQOL-54
Immunology | baseline, month 1
  * Dosing of G, A and M immunoglobulins, and complement factors C3 and C4
  * Determination of lymphocyte subpopulations using cell surface staining and flow cytometry analysis. T lymphocyte subpopulations (CD4 and CD8), B lymphocytes, natural killer (NK) cells, dendritic and T regulatory cells will be analyzed
  * Quantification in serum by "Cytometricbeadarray" (CBA) and subsequent flow cytometry: IL-2, 4, 6, IFN-γ, IL-10, TNF-α or by ELISA: TGF-β and IL-17.
Immunology | baseline, month 3
  * Dosing of G, A and M immunoglobulins, and complement factors C3 and C4
  * Determination of lymphocyte subpopulations using cell surface staining and flow cytometry analysis. T lymphocyte subpopulations (CD4 and CD8), B lymphocytes, NK cells, dendritic and T regulatory cells will be analyzed
  * Quantification in serum by "Cytometricbeadarray" (CBA) and subsequent flow cytometry: IL-2, 4, 6, IFN-γ, IL-10, TNF-α or by ELISA: TGF-β and IL-17.
Axonal effect | baseline, month 12 post-treatment
  - OCT

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramo, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380